CLINICAL TRIAL: NCT03017547
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Preliminary Efficacy Study of IC14 in Acute Respiratory Distress Syndrome
Brief Title: A Phase 2 Study of IC14 in Acute Respiratory Distress Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: seeking funding
Sponsor: Implicit Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AACTT01
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2025-08-20 (Actual); Status verified 2018-05

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IC14 (Experimental): IC14 4 mg/kg IV on Study Day 1, then IC14 2 mg/kg IV once daily on Study Days 2-4.
  Interventions: Drug: IC14
- Placebo (Placebo Comparator): Placebo IV once daily on Study Day 1-4
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IC14 — Blocks CD14 signalling which is responsible for disease pathogenesis in ARDS
  Other Names: monoclonal antibody against CD14
  Arms: IC14
Other: Placebo — sterile normal saline for infusion
  Arms: Placebo

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) patients will be randomized to receive either IC14 (a single dose of 4 mg/kg followed by 2 mg/kg on Days 2-4) or placebo. Study participation will be for a total of 28 days.

DETAILED DESCRIPTION:
Up to 160 patients with ARDS will be randomized to receive either IC14 at a dosage of 4 mg/kg on Study Day 1, then 2 mg/kg once daily on Study Days 2-4 or placebo for 4 days beginning within 48 hours of meeting inclusion criteria. Study participation will be for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. ICU admission
2. Age 18-70 years
3. Presence of a known ARDS clinical risk within 7 days of onset:

   1. Pneumonia
   2. Sepsis
   3. Trauma
   4. Aspiration
   5. Pancreatitis
4. Presence of ARDS (per Berlin criteria) defined as follows:

   1. Acute onset (<48 hours)
   2. PaO2/FiO2<300 on PEEP≥5
   3. Bilateral opacities consistent with pulmonary edema on frontal chest radiograph not fully explained by effusions, lobar/lung collapse, or nodules.
   4. Requirement for positive pressure ventilation via endotracheal tube
5. Anticipated duration of mechanical ventilation >48 hrs

Exclusion Criteria:

1. Treatment with a drug or device within the last 30 days that has not received regulatory approval at the time of study entry
2. Intubation for cardiopulmonary arrest
3. Do-not-attempt resuscitation (DNAR) status
4. Intubation for status asthmaticus, pulmonary embolus, myocardial infarction
5. Anticipated survival <48 hours from intubation
6. Anticipated survival <28 days due to pre-existing medical condition
7. Significant pre-existing organ dysfunction

   1. Lung: Currently receiving home oxygen therapy as documented in medical record
   2. Heart: Pre-existing congestive heart failure defined as an ejection fraction <20% as documented in the medical record
   3. Renal: Chronic renal failure requiring renal replacement therapy
   4. Liver: Severe chronic liver disease defined as Child-Pugh Class C
8. Pre-existing, ongoing immunosuppression

   1. Solid organ transplant recipient
   2. Chronic high-dose corticosteroids (equivalent to >20 mg/prednisone/day for >14 days in the last 30 days)
   3. Oncolytic drug therapy within the past 14 days
   4. Known HIV positive with CD4 count <200 cells/mm3
9. Current treatment with Enbrel® (etanercept), Remicade® (infliximab), Humira® (adalimumab), Cimzia® (certolizumab), or Simponi® (golimumab), Kineret® (anakinra), or Arcalyst® (rilonacept)
10. Pregnancy
11. History of hypersensitivity or idiosyncratic reaction to IC14
12. Deprivation of freedom by administrative or court order

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Safety | 28 days
  Treatment-emergent adverse events
Ventilator-free days | 28 days
  The number of days alive and free of mechanical ventilation through Day 28.

SECONDARY OUTCOMES:
Change in ARDS biologic markers. | 28 days
  * Change in plasma IL-8, sTNFR1, IL-6 from Day 0 to Day 4
  * Change in alveolar neutrophils and total protein from Day 0 to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Jan Agosti, MD, Study Director — Implicit Bioscience